CLINICAL TRIAL: NCT03803774
Title: Birinapant and Intensity Modulated Re-Irradiation Therapy (IMRRT) for Locoregionally Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Birinapant and Intensity Modulated Re-Irradiation Therapy in Treating Patients With Locally Recurrent Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00175; NCI-2019-00175 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-C-0041; 10184 (Other: National Cancer Institute LAO); 10184 (Other: CTEP); NCT03809208 (obsolete NCT alias)
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: Locally Recurrent Head and Neck Squamous Cell Carcinoma; Nasopharyngeal Squamous Cell Carcinoma; Sinonasal Squamous Cell Carcinoma
MeSH Terms: interventions — Biopsy; birinapant; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (IMRRT, birinapant) (Experimental): Beginning on day 1, patients undergo IMRRT 5 days a week (Monday-Friday). Patients also receive birinapant IV over 30 minutes on days 2 and 9 of each cycle. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Drug: Birinapant; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Drug: Birinapant — Given IV
  Other Names: TL32711
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of birinapant when given together with intensity modulated re-irradiation therapy (IMRRT) in treating patients with head and neck squamous cell carcinoma that has come back at or near the same place as the original (primary) tumor (locally recurrent). Birinapant may stop the growth of tumor cells by blocking inhibitor of apoptosis (IAP), a protein needed for tumor cell survival. IMRRT uses thin beams of radiation of different intensities that are aimed at the tumor from many angles. This type of re-irradiation therapy reduces the damage to healthy tissue near the tumor. Giving birinapant with IMRRT may lower the chance of head and neck squamous cell carcinoma growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the toxicities and maximum tolerated dose (MTD) of birinapant concurrent with intensity modulated re-irradiation therapy (IMRRT).

SECONDARY OBJECTIVES:

I. Determine the objective response rate of patients with locoregionally recurrent head and neck squamous cell carcinoma (HNSCC) treated with re-irradiation and birinapant.

II. Determine the local-regional control, progression free survival (PFS), and overall survival.

III. Determine if Fas-associated death domain (FADD) and/or Baculoviral IAP Repeat containing 2 and Baculoviral IAP Repeat containing 3 (BIRC2/3) copy gain in tumor tissue or in the blood are associated with improved response, locoregional control (LCR), progression-free survival and overall survival.

IV. Determine the feasibility of detecting effects of birinapant and re-irradiation on pilot pharmacodynamic markers in tumor tissue, by using microwestern to assess decrease in drug targets inhibitor of apoptosis 1/2 (IAP1/2) and increase in apoptosis/necroptosis markers caspase 3 and mixed lineage kinase domain like pseudokinase gene (MLKL).

EXPLORATORY OBJECTIVES:

I. Explore if mutational load detected with whole exome sequencing of tumor tissue influences objective response rate.

II. Explore if programmed death-ligand 1 (PD-L1), cluster of differentiation 8 (CD8) T-cell tumor infiltration, TNFalphatumor necrosis factor (TNF)alpha, and other immune related biomarkers in tumor tissue are associated with objective response rate.

III. Explore the pharmacokinetics of birinapant in combination with radiotherapy in blood samples.

IV. Explore whether specific germline single-nucleotide polymorphisms (SNPs) are associated with response to birinapant and reirradiation.

OUTLINE: This is a dose-escalation study of birinapant.

Beginning on day 1, patients undergo IMRRT 5 days a week (Monday-Friday). Patients also receive birinapant intravenously (IV) over 30 minutes on days 2 and 9 of each cycle. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days, and at 3, 6, 9, 12, 18, and 24 months until confirmation of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally recurrent HNSCC, including nasopharyngeal or sinonasal cancer for whom re-irradiation for local control is considered standard of care
* Patients with human papillomavirus (HPV)-negative or HPV-positive head and neck cancer are eligible
* Patients who have had prior treatment with immune therapies are eligible
* Patients must have received curative-intent platinum- and/or cetuximab-based chemoradiotherapy or radiotherapy alone
* Patients must have completed their last treatment dose with chemotherapy or immunotherapy at least 4 weeks (6 weeks for nitrosoureas or mitomycin C) before enrolling on study
* Patients must have completed their last treatment dose with radiotherapy at least 6 months before enrolling on study
* Patients who have had major surgery must be fully recovered and require a recovery period of at least 4 weeks prior to enrolling on study
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 9 g/dL (transfusion permitted)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within 1.5 x the upper limit of normal (ULN) institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine =< 1.5 x upper limit of normal (ULN), OR: Creatinine clearance >= 50 mL/min according to Cockcroft Gault formula or other institutional methods
* Patients must have a corrected QT interval by Fridericia (QTcF) =< 480 msec
* International normalized ratio (INR) =< 1.5 and no clinically significant bleeding event within the past six months
* Ability to understand and the willingness to sign a written informed consent document
* Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* The effects of birinapant on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) beginning at study entry and for the duration of study participation. Male study participants should use an additional barrier method of contraception for 30 days following the last dose of birinapant. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Eligibility for curative-intent surgery, unless the patient is considered a poor surgical candidate related to resectability, functional outcome, or prefers non-surgical therapy
* More than 2 lines of palliative systemic therapy (platinum-, taxane- or cetuximab-based chemotherapy or immunotherapy)
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to birinapant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because birinapant may have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with birinapant, breastfeeding should be discontinued prior to enrollment. A negative pregnancy test is required for women of childbearing potential. Women who are postmenopausal (age-related amenorrhea >= 12 consecutive months, or who had undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing. If necessary, to confirm postmenopausal status, a follicle stimulating hormone (FSH) level may be included at screening
* Human immunodeficiency virus (HIV) positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with birinapant
* Patients requiring the use of anti-tumor necrosis factor (anti TNF) therapies, such as infliximab, or patients who have received treatment with anti-TNF therapies within 5 half-lives of the drug (48 days for infliximab, 55 days for golimumab, 70 days for certolizumab and adalimumab, and 16 days for etanercept)
* Patients with previous exposure to birinapant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2026-07-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Saloura, Principal Investigator — National Cancer Institute LAO
Locations (33):
- United States (33):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Birinapant 2.8 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy): SG1 Dose Level -1 Dose Escalation: Up to 24 participants with locally recurrent head and neck squamous cell carcinoma (HNSCC) to determine maximum tolerated dose (MTD) (dose escalation group).
  LEVEL -1: Cycle 1-2 Birinapant 2.8 mg/m^2 intravenous (IV) days 2 & 9; intensity modulated re-irradiation therapy (IMRRT) 2 Gray (Gy) Fx day(d)1-5 every week (QW) for 3 weeks (wk)
- Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy): SG1 Dose Level 1 Dose Escalation: Up to 24 participants with locally recurrent head and neck squamous cell carcinoma (HNSCC) to determine maximum tolerated dose (MTD) (dose escalation group).
  LEVEL 1: Cycle 1-2 Birinapant 5.6 mg/m^2 intravenous (IV) days 2 & 9; intensity modulated re-irradiation therapy (IMRRT) 2 Gray (Gy) Fx day(d)1-5 every week (QW) for 3 weeks (wk)
- Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy): SG1 Dose Level 2 Dose Escalation: Up to 24 participants with locally recurrent head and neck squamous cell carcinoma (HNSCC) to determine maximum tolerated dose (MTD) (dose escalation group).
  LEVEL 2: Cycle 1-2 Birinapant 11 mg/m^2 intravenous (IV) days 2 & 9; intensity modulated re-irradiation therapy (IMRRT) 2 Gray (Gy) Fx day(d)1-5 every week (QW) for 3 weeks (wk)
- Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy): SG1 Dose Level 3 Dose Escalation: Up to 24 participants with locally recurrent head and neck squamous cell carcinoma (HNSCC) to determine maximum tolerated dose (MTD) (dose escalation group).
  LEVEL 3: Cycle 1-2 Birinapant 17 mg/m^2 intravenous (IV) days 2 & 9; intensity modulated re-irradiation therapy (IMRRT) 2 Gray (Gy) Fx day(d)1-5 every week (QW) for 3 weeks (wk)
- Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy): SG1 Dose Level Dose Escalation: Up to 24 participants with locally recurrent head and neck squamous cell carcinoma (HNSCC) to determine maximum tolerated dose (MTD) (dose escalation group).
  Cycle 1-2 Birinapant 24 mg/m^2 intravenous (IV) days 2 & 9; intensity modulated re-irradiation therapy (IMRRT) 2 Gray (Gy) Fx day(d)1-5 every week (QW) for 3 weeks (wk)
Period: Dose Escalation
Arm/Group | Birinapant 2.8 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy)
Started | 0 | 3 | 3 | 4 | 3
Completed | 0 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Dose Expansion
Arm/Group | Birinapant 2.8 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy)
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 1 | 10
  >=65 years | 0 | 0 | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 51.33 [46 to 54] | 55.67 [46 to 62] | 63 [53 to 76] | 71 [63 to 78] | 60.46 [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 2
  Male | 2 | 3 | 4 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 1 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 1 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) and Grades 1-5 Serious and/or Non-serious Toxicities Related (Except for Unrelated and Unlikely) to Intervention
Description: Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. A DLT is defined as any of the following adverse events possibly attributed to the combination of birinapant and radiotherapy that occur within 42 days after treatment. Any grade 5 toxicities. Any grade ≥ 4 hematologic toxicity, except lymphopenia. Any grade ≥ 3 non-hematologic toxicity except for nausea or vomiting managed with supportive care over 2 weeks. ≥ grade 3 prolonged (> 7 days) serum amylase or lipase elevation, aspartate aminotransferase elevation, and/or alanine aminotransferase elevation. Any grade toxicity that mandates discontinuation of birinapant treatment for more than 2 weeks. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Up to 42 days post-treatment
Measure: Number; unit: toxicities
Arm/Group | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy)
Number analyzed (Participants) | 3 | 3 | 4 | 3
toxicities
  Grades 1-5 Dose Limiting Toxicities | 0 | 0 | 0 | 0
  All serious and non-serious Grades 1-5 related adverse events | 66 | 49 | 26 | 1
  All serious Grades 1-5 related adverse events | 2 | 2 | 0 | 1
  Grades 3-5 serious and non-serious related adverse events | 8 | 6 | 3 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Birinapant
Description: MTD is defined as the dose level at which no more than 1 of up to 6 participants experience dose limiting- toxicity (DLT) during 42 days after the start of therapy, and the dose below that at which at least 2 (of =< 6) participants have DLT as a result of the drug. A DLT is defined as any of the following adverse events possibly attributed to the combination of birinapant and radiotherapy that occur within 42 days after treatment. Any grade 5 toxicities. Any grade ≥ 4 hematologic toxicity except lymphopenia. Any grade ≥ 3 non-hematologic toxicity except for nausea or vomiting managed with supportive care over 2 weeks. ≥ grade 3 prolonged (> 7 days) serum amylase or lipase elevation, aspartate aminotransferase elevation, and/or alanine aminotransferase elevation. Any grade toxicity that mandates discontinuation of birinapant treatment for more than 2 weeks. Adverse events were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 42 days
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received birinapant intravenous (IV) over 30 minutes on days 2 and 9 of each cycle. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Participants
Number analyzed (Participants) | 13
mg/m^2 | 24

3. Secondary Outcome: Response Rate
Description: Overall response is the best response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Estimates of response rates will be determined at the maximum tolerated dose (MTD) level, including the expansion cohort and will be presented along with a 95% two-sided confidence interval. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesion. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions; and the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From the start of the treatment until response assessment by positron emission tomography (PET)-computed tomography (CT), assessed at 3 months post-treatment
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Local-regional Control
Description: Estimates of local control will be determined at the maximum tolerated dose (MTD) level, including the expansion cohort and will be presented along with a 95% two-sided confidence interval.
Time Frame: Up to 24 months post-treatment
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Estimates of PFS will be determined at the maximum tolerated dose (MTD) level, including the expansion cohort and will be presented along with a 95% two-sided confidence interval. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions; and the appearance of one or more new lesions.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 24 months post-treatment
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Overall Survival (OS)
Description: OS is the time between the first day of treatment to the day of death. Estimates of OS will be determined at the maximum tolerated dose (MTD) level, including the expansion cohort, and will be presented along with a 95% two-sided confidence interval.
Time Frame: Up to 24 months post-treatment
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Fas-associated Protein With Death Domain (FADD) Copy Gain in Tumor Tissue and/or in Blood Associated With Response
Description: The association between FADD copy gain in tumor tissue and/or in blood will be evaluated for any association with response.
Time Frame: At baseline
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: BIRC2 Copy Gain in Tumor Tissue and/or in Blood Associated With Response
Description: BIRC2 copy gain in tumor tissue and/or in blood will be evaluated for any association with response.
Time Frame: At baseline
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Baculoviral Inhibitor of Apoptosis (IAP) Repeat Containing 2 and Baculoviral IAP Repeat Containing 2/3 (BIRC2/3) Copy Gain in Tumor Tissue and/or in Blood
Description: Baculoviral inhibitor of apoptosis (IAP) Repeat containing 2 and Baculoviral IAP Repeat containing 2/3 (BIRC2/3) copy gain in tumor tissue and/or in blood.
Time Frame: At baseline
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Feasibility of Detecting Effects of Birinapant and Re-irradiation on Pilot Pharmacodynamic Markers in Tumor Tissue
Description: Will determine the feasibility of detecting effects of birinapant and re-irradiation on pilot pharmacodynamic markers in tumor tissue.
Time Frame: Up to cycle 1, day 4
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Feasibility of Detecting Effects of Birinapant and Re-irradiation on Pilot Pharmacodynamic Markers Microwestern for Decrease in Drug Targets Inhibitor of Apoptosis 1/2 (IAP1/2)
Description: Will determine the feasibility of detecting effects of birinapant and re-irradiation on pilot pharmacodynamic markers microwestern for decrease in drug targets IAP1/2.
Time Frame: Up to cycle 1, day 4
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Change in Caspase 3 Levels
Description: A change (i.e., increase) in apoptosis/necroptosis marker caspase 3 will be evaluated.
Time Frame: Baseline up to cycle 1, day 4
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Change in Mixed Lineage Kinase Domain-like (MLKL) Levels
Description: A change (i.e., increase) in apoptosis/necroptosis marker mixed lineage kinase domain-like (MLKL) levels will be evaluated.
Time Frame: Baseline up to cycle 1, day 4
Reporting Status: Not Posted, anticipated posting 2026-03

14. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: An average of 611 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy)
Number analyzed (Participants) | 3 | 3 | 4 | 3
Participants | 3 | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: An average of 611 days.
Arm/Group | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=4) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Iron deficiency anemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vascular disorders - Other, Carotid Occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Birinapant 5.6 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3) | Birinapant 11 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3) | Birinapant 17 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=4) | Birinapant 24 mg/m^2 & Intensity Modulated Re-Irradiation Therapy (IMRRT) 2 Gray(Gy) (N=3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, Blood Clots (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (3) | 3 (6) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, Ear Fullness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5) | 1 (4) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (8) | 3 (4) | 2 (6) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (4) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Neck Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Nerve pain- cheeks (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Neck edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin rash, small red dots chest and abdomen (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03803774/Prot_SAP_000.pdf